CLINICAL TRIAL: NCT06316050
Title: Retrovertion Assesment and Study of the Subscapularis Function in Elderly Patients With Reverse Total Shoulder Arthroplasty
Brief Title: Retrovertion Assesment and Study in Elderly Patients With Reverse Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Josep Maria Mora Guix, Chief of Shoulder Unit, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cst
Record Dates: First submitted 2024-01-16; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Open randomized controlled clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- humeral retroversion 0º (Active Comparator): will be carried out with patients operated with reverse shoulder arthroplasty (at 0º and 30º of humeral retroversion) included consecutively in Terrassa Hospital
  Interventions: Procedure: humeral retroversion
- humeral retroversion 30º (No Intervention): will be carried out with patients operated with reverse shoulder arthroplasty (at 0º and 30º of humeral retroversion) included consecutively in Terrassa Hospital

INTERVENTIONS:
Procedure: humeral retroversion — REVERSED SHOULDER ARTHROPLASTY IN TWO DIFFERENT GROUPS. Group 0 humeral retroversion, Group 30º humeral retroversion
  Arms: humeral retroversion 0º

SUMMARY:
Determine the optimal degree of retroversion (0-30º) to obtain the best rotational mobility, both internal and external, of the shoulder after implanting a reversed sghoulder arthroplasty (Comprehensive system), and analyze the functional and radiologic results based on humeral retroversion.

DETAILED DESCRIPTION:
Methodology: Open randomized controlled clinical trial. It will be carried out with patients operated with reverse shoulder arthroplasty (at 0º and 30º of humeral retroversion) included consecutively in Terrassa Hospital from January 2019 to June 2021. The estimated sample will be 30 patients per group with diagnosis of massive rotator cuff rupture, rotator cuff arthropaty and primary osteoarthritis with cuff injury, with Walch's type B2 glena or in patients older than 80 years. A global study will be carried out preoperatively and postoperatively with radiographs, computerized tomography, magnetic resonance, and a biomechanical study.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 60 with the diagnosis rotator cuff massive break (Hamada 2 or more), arthrosis secondary to ruptures of the rotator cuff and primary osteoarthritis with lesion of the cuff, with full Walch B2 type or in patients older than 80 years. Inclusion criteria
* Good functionality of the deltoid muscle.
* Presence of minor round (Hornblower test - no muscle atrophy in nuclear magnetic resonance)
* Accept informed consent

Exclusion Criteria:

* - Review of hemiarthroplasty or anatomical proesis of the affected shoulder.
* Fracture of shoulder in the upper extremity to intervene.
* Central neurological diseases
* Advanced cognitive impairment
* Brachial plexus injuries
* Local or systemic infection.
* Oncological disease
* Treatment with immunosuppressants.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
INTERNAL ROTATION | 2 YEARS
  AT THE SIDE (HAND TO the BACK from CONSTANT TEST)
INTERNAL ROTATION | 2 YEARS
  degrees

SECONDARY OUTCOMES:
EXTERNAL ROTATION | 2 YEARS
  degrees
FORWARD ELEVATION | 2 YEARS
  degrees
Simple shoulder test | 2 years
  0-100
Constant test | 2 years
  0-100
ASES test | 2 years
  0-100
Glenoid inclination angle | 2 years
  degrees
glenoid retroversion angle | 2 years
  degrees
abduction | 2 years
  degrees
center of rotation | 2 years
  milimiters
lateralizaiton offset | 2 years
  milimiters

CONTACTS AND LOCATIONS:
Locations (1):
- JM MORA, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR